CLINICAL TRIAL: NCT01720212
Title: An Open-Label, Single and Multiple Dose Study to Assess the Safety and Pharmacokinetics of YM178 OCAS Tablet (Mirabegron) in Healthy Chinese Volunteers
Brief Title: Study to Assess the Safety and Plasma Concentration of YM178 OCAS Tablet (Mirabegron) in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 178-CL-091
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Chinese Volunteers
Keywords: YM178; Mirabegron; OCAS; Chinese Healthy Volunteers; PK; Safety
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose group (Experimental)
  Interventions: Drug: YM178
- Multiple dose group (Experimental)
  Interventions: Drug: YM178

INTERVENTIONS:
Drug: YM178 — oral
  Other Names: Mirabegron

SUMMARY:
To evaluate the safety and plasma concentration change of YM178 after single- and repeated-administration as oral absorption controlled tablet in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) between 19 and 24, the weight is no less than 50 kg.
2. Good health status
3. The female subject must be either post-menopausal or surgically sterile. All women of child bearing potential will be required to use adequate contraception, must not be lactating, and must not be breastfeeding.

Exclusion Criteria:

1. The subject who has a known or suspected hypersensitivity to test drug or any of the constituents of the formulation used.
2. Drug abusers and alcoholics.
3. The subject who has consumed alcohol within 36 hours before administration.
4. The subject who is positive for hepatitis B surface antigen (HBs- Ag) or hepatitis C virus (HCV) antibody.
5. The subject who is positive for human immunodeficiency virus (HIV).
6. The subject who consumes more than 1L tea and coffee per day.
7. Smokers.
8. The subject who has donated or lost over 200 mL blood
9. The subject who has participated in other clinical trials
10. The subject who has taken other drugs that prototype and its main metabolites had not completely eliminated
11. The subject who has taken drugs repeatedly that may affect the metabolism of the test drug
12. Psychopath.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
AUC of YM178 assessed by the plasma concentration changes | Up to 96 hours after administration
Cmax of YM178 assessed by the plasma concentration changes | Up to 96 hours after administration
t1/2 of YM178 assessed by the plasma concentration changes | Up to 96 hours after administration

SECONDARY OUTCOMES:
Safety assessment of YM178 | Up to 33 days
  Safety is to be assessed by the incidence of adverse events, vital signs, lab-tests and 12-lead ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Shanghai, China